CLINICAL TRIAL: NCT04387552
Title: Improving Care Giver Adherence to Recommended Infant Care Practices
Brief Title: Social Media and Risk Reduction Teaching-Enhanced Reach
Acronym: SMARTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: University of Virginia (Other); Washington University School of Medicine (Other); Boston Medical Center (Other); University of Kentucky (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: H-39495; R01HD072815-06A1 (NIH)
Record Dates: First submitted 2020-05-10; First posted 2020-05-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breastfeeding; SUID; SIDS
Keywords: Breastfeeding (BF); Sleep position; Safe Sleep (SS); Mobile Messaging; Social Media; WIC
MeSH Terms: conditions — Breast Feeding; Sudden Infant Death | interventions — Telemedicine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prenatal SS/Postnatal BF (Experimental): Prenatal Safe Sleep/Postnatal Breastfeeding Mobile Health Messages
  Interventions: Behavioral: Prenatal Safe Sleep Mobile Health (mHealth) Messaging; Behavioral: Postnatal Breastfeeding Mobile Health (mHealth) Messaging
- Prenatal BF/Postnatal SS (Experimental): Prenatal Breastfeeding/Postnatal Safe Sleep Mobile Health Messages
  Interventions: Behavioral: Prenatal Breastfeeding Mobile Health (mHealth) Messaging; Behavioral: Postnatal Safe Sleep Mobile Health (mHealth) Messaging
- Prenatal SS/Postnatal SS (Experimental): Prenatal Safe Sleep/Postnatal Safe Sleep Mobile Health Messages
  Interventions: Behavioral: Prenatal Safe Sleep Mobile Health (mHealth) Messaging; Behavioral: Postnatal Safe Sleep Mobile Health (mHealth) Messaging
- Prenatal BF/Postnatal BF (Experimental): Prenatal Breastfeeding/Postnatal Breastfeeding Mobile Health Messages
  Interventions: Behavioral: Prenatal Breastfeeding Mobile Health (mHealth) Messaging; Behavioral: Postnatal Breastfeeding Mobile Health (mHealth) Messaging

INTERVENTIONS:
Behavioral: Prenatal Safe Sleep Mobile Health (mHealth) Messaging — Participants will receive prenatal Safe Sleep mHealth messaging starting at 34 weeks gestation until birth of their baby.
  Arms: Prenatal SS/Postnatal BF; Prenatal SS/Postnatal SS
Behavioral: Prenatal Breastfeeding Mobile Health (mHealth) Messaging — Participants will receive prenatal Breastfeeding mHealth messaging starting at 34 weeks gestation until birth of their baby.
  Arms: Prenatal BF/Postnatal BF; Prenatal BF/Postnatal SS
Behavioral: Postnatal Safe Sleep Mobile Health (mHealth) Messaging — Upon birth of baby, participants will begin receiving postnatal Safe Sleep mHealth messaging for a two month period.
  Arms: Prenatal BF/Postnatal SS; Prenatal SS/Postnatal SS
Behavioral: Postnatal Breastfeeding Mobile Health (mHealth) Messaging — Upon birth of baby, participants will begin receiving postnatal Breastfeeding mHealth messaging for a two month period.
  Arms: Prenatal BF/Postnatal BF; Prenatal SS/Postnatal BF

SUMMARY:
This study aims to improve adherence to American Academy of Pediatrics safe sleep (SS) recommendations and improve rates of initiation and duration of partial and exclusive breastfeeding (BF) through direct education of mothers using Mobile Health (mHealth) technologies (ex. text messaging).

DETAILED DESCRIPTION:
The goal of this study is to assess the effectiveness of mHealth prenatal and postnatal interventions aimed at promoting safe sleep (SS) practices and breastfeeding (BF) within a population of pregnant Supplemental Nutrition Program for Women, Infants, and Children (WIC) clients.

The study will randomize 2,000 pregnant women, when they reach 34 weeks gestation, to one of four mHealth prenatal/postnatal messaging combinations of safe sleep and breastfeeding practices.

ELIGIBILITY:
Inclusion Criteria:

* Must be client at a WIC center participating in study.
* Must be pregnant and less than 34 weeks gestation
* Must speak English or Spanish
* Must live in the United States
* Must have texting capabilities via mobile phone
* Must plan to live in same household as infant after birth.

Exclusion Criteria:

* A prenatal diagnosis expected to have impact on infant care practices not compatible with study goals, including contraindications to breastfeeding or supine infant sleep positioning.
* Meets the definition of a minor according to applicable state law.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2126 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2025-06-07 (Actual); Study Completion 2025-06-07 (Actual)

PRIMARY OUTCOMES:
Infant sleep position in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess infant's sleep position during the previous two weeks with categorical responses of back, stomach, side, and other. We will examine: A) Usual position; B) Exclusive use of supine position
Infant sleep location in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess the infant's sleep location during the previous two weeks with categorical responses of room sharing without bed sharing, room sharing with bed sharing, no room sharing and no bed sharing. We will examine: A) Usual location; B) Exclusive location of room sharing without bedsharing
Any Soft bedding use in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess soft bedding placed in and around the infant (while sleeping) during the previous two weeks with categorical responses of Yes or No.
Any Pacifier use in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess the infant's pacifier use during the previous two weeks with categorical responses of Yes or No.
Infant feeding in the previous two weeks | Between 2 and 6 months
  An investigator-developed maternal survey will be used to assess whether the infant was breast fed during the previous two weeks with categorical responses of exclusively breast fed, partially breast fed, or not breast fed. We will examine: A) Any breast milk feeding; B) Exclusive breast milk feeding

SECONDARY OUTCOMES:
Any Initiation of breast milk feeding | Between 36 weeks gestational age and birth
  The impact of the only the prenatal intervention on initiation of breast milk feeding obtained through maternal survey responses on the prenatal survey
Planned infant sleep position after birth of baby | Between 36 weeks gestational age and birth.
  The impact of the only the prenatal intervention on planned infant sleep position after birth of baby obtained through maternal survey responses on the prenatal survey
Planned infant sleep location after birth of baby | Between 36 weeks gestational age and birth.
  The impact of the only the prenatal intervention on planned infant sleep location after birth of baby obtained through maternal survey responses on the prenatal survey
Planned breast milk feeding after birth of baby | Between 36 weeks gestational age and birth.
  The impact of the only the prenatal intervention on planned breast milk feeding after birth of baby obtained through maternal survey responses on the prenatal survey
Planned duration of breast milk feeding after birth of baby | Between 36 weeks gestational age and birth
  An investigator-developed maternal prenatal survey will be used to assess planned duration of breast milk feeding after birth of baby obtained through maternal survey responses on the prenatal survey
Days from postnatal randomization to first report of not exclusively in the supine sleep position | Weekly until the infant is 26 weeks of age.
  The number of days after postnatal randomization when supine sleep position is stopped will be assessed by maternal response to weekly text messages about sleep position during the past week.
Days from postnatal randomization to first report of not exclusively room sharing without bed sharing | Weekly until the infant is 26 weeks of age.
  The number of days after postnatal randomization when sleep location of room sharing without bed sharing stopped will be assessed by maternal response to weekly text messages about sleep location during the past week.
Days from postnatal randomization to first report of using any soft bedding | Weekly until the infant is 26 weeks of age.
  The number of days after postnatal randomization when soft bedding use starts will be assessed by maternal response to weekly text messages about type of bedding during the past week.
Days from postnatal randomization to first report of not receiving exclusively Breast Milk feedings | Weekly until the infant is 26 weeks of age.
  The days from postnatal randomization when breast feeding changed will be assessed by maternal response to weekly text messages about type of breast feeding categorized as either exclusive, partial or no breast milk during the past week.
Days from postnatal randomization to first report of not receiving any Breast Milk feedings | Weekly until the infant is 26 weeks of age.
  The number of days after postnatal randomization to first report of not receiving any Breast Milk feedings will be assessed by maternal response to weekly text messages about type of breast feeding categorized as or no breast milk during the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Corwin, MD, Principal Investigator — Boston University School of Public Health, Dept of Pediatrics, BUSM
Locations (1):
- Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No